CLINICAL TRIAL: NCT04332562
Title: The Association Between Serum β-hydroxybutyrate and Levels of Systemic Hypertension: "An Open-label Randomized Controlled Trial.
Brief Title: The Association Between Serum β-hydroxybutyrate and Levels of Systemic Hypertension
Acronym: BHB-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sulaiman AlRajhi Colleges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SulaimanAC- BHB
Record Dates: First submitted 2020-01-20; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Hypertension, Essential; β-hydroxybutyrate
Keywords: β-hydroxybutyrate; Hypertension
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normotensive control group (No Intervention): Normotensive volunteer
- hypertensive control group (No Intervention): Hypertensive patients with no restriction on their salt intake
- hypertensive interventional group (Experimental): intervention is going to be salt restriction
  Interventions: Other: dietary restriction (salt restriction)

INTERVENTIONS:
Other: dietary restriction (salt restriction) — salt restriction for one week after being diagnosed with hypertension
  Arms: hypertensive interventional group

SUMMARY:
In this research the investigators are looking for the direct relationship between Beta-hydroxybutyrate and hypertension. Since recent research showed a connection between exercise and hypertension, and diet control and hypertension. The investigators are studying the possible effect of beta-hydroxybutyrate levels on blood pressure control.

DETAILED DESCRIPTION:
Systemic hypertension is defined as a systolic blood pressure that is ≥ 140 mm hg and / or a diastolic blood pressure that is ≥ 90 mm hg a modifiable and it is known to be a serious risk factor for cardiovascular disease. Exercise is widely recommended as a lifestyle modification for hypertensive patients because of its beneficial effect on lowering blood pressure (BP). Similarly, calorie restriction is also documented to lower systemic hypertension.

Interestingly, both exercise and calorie-restriction are associated with increased circulating levels of ketone bodies such as β-hydroxybutyrate (βHB). β-Hydroxybutyrate (βHB; 3-hydroxybutyric acid) is a "ketone body" which is produced the liver, mainly from the oxidation of fatty acids, and is exported to peripheral tissues for use as an energy source. It is transported to extrahepatic tissues, and traditionally recognized as a vital alternative source of energy during starvation. However, recent evidences indicate that apart from serving as energy fuel, ketone bodies such as βHB block nucleotide-binding domain, leucine-rich-containing family, pyrin domain-containing-3 (Nlrp3)-inflammasome-mediated inflammatory diseases, and thereby play a prominent role in maintaining physiological homeostasis parameter such as blood pressure.

Among environmental factors, excessive salt intake is the most common and important risk factor for hypertension, in which patient with salt-sensitive hypertension demonstrated an increased risk of cardiovascular disease. There is substantial evidence suggesting that blood pressure's (BP) response to dietary salt intake vary considerably among individuals which is a phenomenon described as salt sensitivity of blood pressure.

Another reference demonstrated a lower circulating level of the ketone body, beta-hydroxybutyrate (βHB), in high salt-fed hypertensive rats. Despite the high salt intake, the specific rescue of (βHB) levels by nutritional supplementation of its precursor, 1,3-butanediol, attenuates hypertension and protects kidney function by inhibiting the renal Nlrp3 inflammasome in rats.

Existing Knowledge and Literature Review: PubMed search builder was used to construct the following search entry: hypertension AND β-Hydroxybutyrate. The initial search yielded 39 titles. Studies (RCTs or systemic reviews) relevant to the research question were isolated manually by reading the abstracts. However, due to the novelty of the idea, the investigators were not able to identify any related literature except of "Chakraborty, Saroj" study. which was a non-human research.

Research impact: The current evidence regarding the effect of β-Hydroxybutyrate supplementation on the reduction of salt-sensitive hypertension was only proven on a non-human level. The research will address this gap in knowledge by looking for any relationship between the levels of (βHB) and salt-sensitive hypertensive in human subjects, which may change the current understanding of the treatment of salt-sensitive.

ELIGIBILITY:
Inclusion Criteria for:

1. All patients ≥ 18 years
2. not diagnosed with systemic hypertension

Inclusion Criteria for:

1. All patients ≥ 18 years
2. First time diagnosed as a case of systemic hypertension

Exclusion Criteria:

1. Diabetes mellitus.
2. Previous heart diseases, kidney or liver diseases as these conditions may interfere with the serum levels of β-hydroxybutyrate.
3. Patients using diuretics.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-15 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-28 (Estimated)

PRIMARY OUTCOMES:
scanning for levels of circulating βHB mmol/L in the serum of the participant | 1 week
  scanning for levels of circulating βHB in mmol/L in the serum of the hypertensive arm in comparison to the control arm.

SECONDARY OUTCOMES:
The correlation between the salt intake restriction and it is effect on the blood pressure in (mmHg) . | 2 weeks
  Hypertensive participant on salt restriction to under go a serial measurement of their blood pressure ( mmHg) .
The effect of salt intake (restriction) on the serum level of βHB mmol/L. | 2 weeks
  Hypertensive participants on salt intake restriction to under go a serial measures of the serum βHB levels mmol/L , looking for any correlation ( if any ) .

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Sherif, MD, Principal Investigator — Sulaiman AlRajhi Colleges

IPD SHARING:
Plan to Share IPD: No